CLINICAL TRIAL: NCT04676256
Title: Comparaison de la Vitrectomie précoce et de la Surveillance Simple Dans la Prise en Charge Des hémorragies du vitré spontanées EVIDENSE Early VItrectomy in DENse Spontaneous Vitreous HEmorrhage
Brief Title: Early VItrectomy in DENse Spontaneous Vitreous HEmorrhage
Acronym: EVIDENSE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P170408J; IDRCB (Other: 2019-A019556-51)
Record Dates: First submitted 2020-01-31; First posted 2020-12-21 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Spontaneous Vitreous Hemorrhage; Retinal Break; Retinal Detachment
Keywords: spontaneous vitreous hemorrhage; retinal break; retinal detachment; ultrasound; vitrectomy
MeSH Terms: conditions — Retinal Perforations; Retinal Detachment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early Vitrectomy (Experimental): Experimental arm will be treated with early vitrectomy early vitrectomy 7 days after vitreous hemorrhage diagnosis
  Interventions: Procedure: Early vitrectomy
- Comparator (Active Comparator): Active comparator arm will have fundus and ultrasound observation. Late vitrectomy may be indicated after 3 months of follow-up if needed.
  Late vitrectomy will be performed in case of persistant vitreous hemorrhage after 3 months of folllow-up
  Interventions: Procedure: Early vitrectomy

INTERVENTIONS:
Procedure: Early vitrectomy — Eyes with spontaneous vitreous hemorrhage treated with early vitrectomy (n = 63)

SUMMARY:
The aim of the protocol is to compare the ocular outcomes after spontaneous vitreous hemorrhage treated with an early vitrectomy versus ultrasound monitoring with late vitrectomy.

The hypothesis is that an early vitrectomy could decrease the rate of retinal detachment occurring after a spontaneous vitreous hemorrhage.

DETAILED DESCRIPTION:
The aim of the protocol is to compare the ocular outcomes after spontaneous vitreous hemorrhage treated with an early vitrectomy versus ultrasound monitoring with late vitrectomy.

The hypothesis is that an early vitrectomy could decrease the rate of retinal detachment occurring after a spontaneous vitreous hemorrhage.

Scientific background Spontaneous vitreous hemorrhage may occur after spontaneous posterior vitreous detachment and causes retinal break and retinal detachment in about 70% and 40% of cases respectively. The fundus examination and ultrasound have limited sensitivity to detect retinal breaks in these cases. Some retrospective studies have highlighted the benefit of an early vitrectomy for decreasing the rate of visual loss due to retinal detachment in these cases. However, to date, there is no national or international consensus regarding the management of spontaneous vitreous hemorrhage and the timing of vitrectomy.

Study design Prospective randomized clinical trial Primary objective To compare the results of an early vitrectomy versus ultrasound and fundus observation in spontaneous vitreous hemorrhage.

Secondary objectives To evaluate the rate of retinal complications in spontaneous vitreous hemorrhage treated either with early or delayed vitrectomy.

To evaluate the rate of visual loss in spontaneous vitreous hemorrhage treated either with early or delayed vitrectomy.

Primary criteria Rate of retinal detachment in eyes with spontaneous vitreous hemorrhage treated with early vitrectomy versus ultrasound observation at 6-month follow-up Secondary criteria Rate of retinal breaks and vitreo-retinal proliferation in eyes with spontaneous vitreous hemorrhage treated with early vitrectomy versus ultrasound observation at 6-month follow-up Visual acuity and rate of eyes with a loss of 5 letters or more among eyes with spontaneous vitreous hemorrhage treated with early vitrectomy versus ultrasound observation at 6-month follow-up Participants Patients with a spontaneous vitreous hemorrhage secondary to posterior vitreous detachment, with a reduced visibility of the fundus Inclusion criteria

* Age > or = 18 years old
* Spontaneous vitreous hemorrhage which is 1/ secondary to posterior vitreous detachment; 2/ acute: which duration is < 15 days, 3/ dense: reduced visibility of the fundus

Exclusion criteria:

* Retinal detachment at the initial examination
* Any history of vascular retinal disease (diabetic retinopathy, retinal vein occlusion…)
* Any history of uveitis, age-related macular degeneration
* History of a recent ocular traumatism (< 3 months)
* History of a recent retinal laser treatment (< 3 months) or vitreo-retinal surgery (< 3 months)
* Absence of consent Experimental group Eyes with spontaneous vitreous hemorrhage treated with early vitrectomy (n = 63) Active Comparator group Eyes with spontaneous vitreous hemorrhage only observed using fundus examination and B-ultrasound (n = 63) Study duration Inclusion: 12 months Participation: 6 months Total duration: 18 months

ELIGIBILITY:
Inclusion Criteria:

* Age > or = 18 years old
* Spontaneous vitreous hemorrhage which is :

  1. secondary to posterior vitreous detachment;
  2. acute: which duration is < 15 days,
  3. dense: reduced visibility of the fundus

Exclusion Criteria:

* Retinal detachment at the initial examination
* Any history of vascular retinal disease (diabetic retinopathy, retinal vein occlusion…)
* Any history of uveitis, age-related macular degeneration
* History of a recent ocular traumatism (< 3 months)
* History of a recent retinal laser treatment (< 3 months) or vitreo-retinal surgery (< 3 months)
* Absence of oral and written consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2021-07-02 (Actual); Primary Completion 2025-01-02 (Estimated); Study Completion 2025-01-02 (Estimated)

PRIMARY OUTCOMES:
Rate of retinal detachment | 6 months after intervention
  number of eyes with a retinal detachment in each group. The presence of retinal detachment will be assessed on fundus examination

SECONDARY OUTCOMES:
Rate of retinal breaks | 6 months after intervention
  number of eyes with a retinal breaks in each group. The presence of retinal breaks will be assessed on fundus examination
Rate vitreo-retinal proliferation | 6 months after intervention
  number of eyes with a vitreo-retinal proliferation in each group. The presence of vitreo-retinal proliferation will be assessed on fundus examination
Visual acuity | 6 months after intervention
  visual acuity will be measured using Snellen and/or ETDRS chart
Rate of eyes with a loss of 5 letters or more | 6 months after intervention
Rate of cataract | 6 months after intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Lariboisiere, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No